CLINICAL TRIAL: NCT02821299
Title: Clinical Evaluation of Laryngeal Transplantation: Pilot Study of 3 Patients
Brief Title: Clinical Evaluation of Laryngeal Transplantation: Study of 3 Patients
Acronym: ECLAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL14_0443; 2016-A00767-44 (Other: DGS)
Record Dates: First submitted 2016-06-09; First posted 2016-07-01 (Estimated); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Laryngeal Transplantation
Keywords: Laryngeal transplantation; Laryngeal function; Swallowing; Voice production; Respiration; Quality of life
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Laryngeal transplantation (Experimental): Laryngeal transplantation
  Interventions: Other: Laryngeal transplantation

INTERVENTIONS:
Other: Laryngeal transplantation — Laryngeal transplantation

SUMMARY:
The experience of face and hand composite tissue transplantations reported in the international community have mainly concerned trauma patients. Feasibility and individual benefit have been demonstrated for these indications, in properly selected patients. The first laryngeal transplantation also concerned a case of post-traumatic reconstruction. A certain number of patients, who have suffered direct (extended period of intubation during a stay in the ICU, road traffic accident etc.) or indirect trauma (thermal or chemical burns) to the larynx, present irreversible trauma or injury to the larynx in which conventional treatments are unable to restore laryngeal function. These patients find themselves severely disabled, with a significant reduction in their quality of life. They suffer from stigmatization which leads to social isolation (professional and personal). In some circumstances, providing healthy tissue and anatomical or functional components (cartilage, muscle, nerves, blood vessels) by means of an allogeneic laryngeal transplantation, is the only way of allowing patients, whose quality of life has been seriously affected, to speak, breath and swallow normally. The extremely promising results from other international teams in this area have encouraged the investigators to present this project.

The specificities of the protocol compared to previous transplantations carried out by other teams are:

* The technique for nerve re-innervation which should make it possible to decannulate all patients and improve functional outcomes in the graft.
* A dual therapy immunosuppressive regimen will be used, if the patient's clinical and biological status permits, which can be adjusted according to the type of tissue grafted.

It might be thought that the need for immunosuppressive therapy means the indications will remain rare, representing an incidence of less than five patients a year in France. However, the interest of this research project does not reside in the number of patients concerned but rather the total lack of any existing therapeutic solution. Conducting a case series will help determine whether, under certain conditions, laryngeal transplantation can improve the management of patients for whom the usual reconstructive surgery options are unsatisfactory.

The study is intended to provide a descriptive analysis of a case series of three laryngeal transplantations before and after comparisons, each patient serving as their own control.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with the permanent loss of laryngeal functions. Loss of laryngeal function is considered when a patient is permanently tracheotomized, is mutic and presented failure for each of the three conventional treatment. Conventional treatment lines are organized in the following manner firstly laser, then prosthesis and lastly surgery) Diet may be normal.
* Adults aged between 18 to 60 years;
* ASA (American Society of Anesthesiology) score < 3 and the health status of the patients must be compatible not only with the graft but also with all the treatments envisaged by the study (according investigator assessment);
* Psychological maturity: recipients should be psychologically balanced, assessed by the team psychiatrists, have taken personality tests, determined and willing, capable of understanding the information provided on the risks relating to the surgery and the immunosuppressive treatment, and capable of making their own decision regarding the transplantation. The psychological preparation for the transplantation requires relationships to be built up prior to the procedure between the patient, the team providing care for laryngectomized patients, the rehabilitation team, the surgical team and the psychiatrist;
* Patients capable of understanding the information provided on the risks relating to the study, and capable of making their own decision regarding the transplantation according investigator assessment;
* Having given written informed consent prior to any procedure related to the study;
* Covered by a Health System where applicable, and/or in compliance with the recommendations of the national laws in force relating to biomedical research.

Exclusion Criteria:

* Minors or patients aged over 60 years;
* Patients with a history of cancer of the upper airways or upper digestive tract;
* Patients with a history of other types of malignancy;
* Patients presenting with a progressive malignant tumor; suspicious laryngeal lesions (dysplasia ...)
* Patients with addiction to alcohol and/or smoking
* Patient presenting hepatitis B, hepatitis C, or HIV(Human Immunodeficiency Virus) infection;
* Patients with a history of psychiatric disorders: known delusional psychosis, untreated severely depressed patients, patients with severe behavioral disorders, patients with permanent generalized anxiety disorder,
* ASA (American Society of Anesthesiology) score ≥ 3;
* Patients presenting moderate renal failure which does not justify renal transplantation with a glomerular filtration rate of less than 60 mL/min per 1.73 m2 calculated using the CKD-EPI formula;
* Arterial hypertension treated by more than one therapy;
* Testing for anti-HLA antibodies will be carried out at the initial inclusion visit, a cross-match will be carried out immediately before transplantation, a positive cross-match will be considered as an automatic contraindication to carrying out the transplantation;
* Women who are pregnant or not taking contraception (effective contraceptive method compulsory);
* Women who are breastfeeding;
* People who have been deprived of their freedom through a legal or administrative decision;
* Adult with a legal guardian;
* Patients in emergency situations;
* EBV (Epstein-Barr Virus) seronegative recipient with EBV seropositive graft, due to the risk of lymphoma.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Estimated)
Dates: Start 2018-09-20 (Actual); Primary Completion 2030-09-20 (Estimated); Study Completion 2030-09-20 (Estimated)

PRIMARY OUTCOMES:
Swallowing evaluation measured using the "Deglutition Handicap Index" | 3 years post transplantation
  The laryngeal transplantation will be evaluated with a primary composite endpoint based on the three inseparable laryngeal functions: swallowing evaluation will be mainly measured using the "Deglutition Handicap Index"
Voice production evaluated by self-report VHI (Voice Handicap Index) patient questionnaires | 3 years post transplantation
  The laryngeal transplantation will be evaluated with a primary composite endpoint based on the three inseparable laryngeal functions: Voice production will be evaluated by self-report VHI (Voice Handicap Index) patient questionnaires
Respiration evaluated by decannulation | 3 years post transplantation
  The laryngeal transplantation will be evaluated with a primary composite endpoint based on the three inseparable laryngeal functions: Respiration, for which the decannulation remains the most appropriate criterion.
Graft survival | 3 years post transplantation

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Service d'Urologie et Chirurgie de la Transplantation - Hôpital Edouard Herriot - Hospices Civils de Lyon, Lyon
  - Service ORL & Chirurgie Cervicofaciale - Hôpital Charles Nicolle - CHU Rouen, Rouen
  - Centre de soins de suite et de réadaptation fonctionnelle - SSR Val Rosay, Saint-Didier-au-Mont-d'Or